CLINICAL TRIAL: NCT04796376
Title: The Outcome of Combined Partial Fistulectomy or Fistulotomy and Cutting Seton Procedure in High Perianal Fistula: Prospective Study
Brief Title: The Outcome of Combined Partial Fistulectomy or Fistulotomy and Cutting Seton Procedure in High Perianal Fistula
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina Nabil Zaher, Resident at General surgery department, faculty of medicine, Assiut University, Egypt, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AssiutU MNZaher
Record Dates: First submitted 2021-02-19; First posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-02

CONDITIONS: High Anal Fistula
Keywords: Cutting seton; Fistulectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cutting seton (Other): A piece of surgical thread that's left in the fistula for several weeks to keep it open. This allow it to drain and help its heal.
  Interventions: Procedure: combined partial fistulectomy or fistulotomy and cutting seton procedure

INTERVENTIONS:
Procedure: combined partial fistulectomy or fistulotomy and cutting seton procedure — Partial excision of fistulous tract or just fistulotomy plus cutting seton procedure which is a rubber band or threads put through fistulous tract

SUMMARY:
The aim of this study is to assess the effectiveness and suitability of the tight (cutting) seton as a surgical treatment of high anal fistula combined with partial fistulotomy or fistulectomy in a prospective study.

DETAILED DESCRIPTION:
Anal fistula is an abnormal tract with two openings: external one opens in perianal skin and the internal one opens in anal canal. And according to relation between fistula and anal sphincters there are intersphincteric, transphincteric, suprasphincteric and extrasphincteric. Varieties of surgical procedures are encountered for management of this disease but complications such as recurrence and incontinence still facing surgeons strongly. In previous study of total 31 patients post-operative complications were; incontinence of gas (16.13%), incontinence of stool (3.23%), recurrence (3.23%) with conclusion of that: outcomes of fistulotomy with cutting seton were satisfactory in most patients (1). In this study and aiming to reduce the complications rate data will be collected about the outcomes of combined partial fistulectomy or fistulotomy and cutting seton procedure in a prospective study. The goals of treatment are draining infection, eradicating the fistulous tract and avoiding persistent or recurrent disease while preserving anal sphincter function.

ELIGIBILITY:
Inclusion Criteria:

* Adult with age of or above 18 years.
* Patients with high perianal fistula; trans-sphincteric, intra-sphincteric or supra-sphincteric.
* Patients sable to comply to with the study protocol.

Exclusion Criteria:

* Patients with low perianal fistula
* Patients with preoperative incontinence.
* Patients with comorbidities such as TB , malignancy or inflammatory bowel disease.
* Patients diagnosed with acute anal sepsis
* Recurrent cases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-10-10 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
- Cure of high perianal fistulas -Reduce incontinence rate | 1 year
  Cure from the main problem of the patient and prevent its recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Mina Nb Zaher, Resident doc, Principal Investigator
Locations (1):
- Assiut University, Asyut, Egypt